CLINICAL TRIAL: NCT05263271
Title: A Phase Ia, Open-label, Dose Escalation Study of Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of Gentulizumab in Patients With Relapsed/Refractory Acute Myelogenous Leukemia or Myelodysplastic Syndrome
Brief Title: Gentulizumab in Relapsed/Refractory Acute Myelogenous Leukemia or Myelodysplastic Syndrome
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changchun GeneScience Pharmaceutical Co., Ltd. (Industry)
Collaborators: Ruijin Hospital (Other); Shanghai Tong Ren Hospital (Other); First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Gensci059-Ia-B
Record Dates: First submitted 2021-12-24; First posted 2022-03-02 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Acute Myelogenous Leukemia; Myelodysplastic Syndromes
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes

STUDY DESIGN:
Intervention Model Description: Part one, priming dose exploration: 5 dose levels (0.03 mg/kg, 0.1 mg/kg, 0.3 mg/kg, 1 mg/kg, 3 mg/kg) Part two, therapeutic dose exploration: 3 dose levels (10 mg/kg,30 mg/kg,45 mg/kg)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental cohort (Experimental): Gentulizumab administered IV once a week and a dosing cycle is 4 weeks
  Interventions: Drug: Gentulizumab

INTERVENTIONS:
Drug: Gentulizumab — Gentulizumab will be administered by intravenous infusion once a week, with every 28 days as a dosing cycle .

SUMMARY:
Gentulizumab Injection is an anti-CD47 monoclonal antibody. As a member of the immunoglobulin superfamily, CD47 is expressed at low levels on many cells of the body, including hematopoietic cells (red blood cells, lymphocytes, platelets, etc.) and non-hematopoietic cells (placenta, liver and brain cells). It is overexpressed on many types of tumors. There is abundant supportive evidence that the expression of CD47 on tumor cells, though binding to SIRP on professional phagocytes, acts to prevent tumor cell phagocytosis, inhibit antigen cross-presentation, and block the production of pro-inflammatory molecules, thus promoting the development of a "cold" tumor microenvironment. Blocking CD47 can not only stimulate phagocytosis to cancer cells, but also promote macrophage recruitment towards neoplasm. At the same time, blocking CD47 can stimulate macrophages to secrete cytokines. These cytokines and chemokines can further recruit other immune cells to neoplasms. These newly recruited immune cells can provide a positive feedback and enhance the therapeutic response of blocking CD47. Therefore, the CD47/SIRPα axis blocking appears to be a potential therapeutic target for neoplasm.

Currently, no anti-CD47 antibody product has been granted marketing authorization for progressive hematological malignancies. Whereas Hu5F9-G4, a CD47 monoclonal antibody, is being tested in a series of ongoing clinical trials for AML, MDS, lymphomas and multiple solid tumors. The clinical research was designed based on non-clinical data and relevant experience of other CD47 monoclonal antibody.

In this phase Ia study, "3 + 3" dose escalation method combined with rapid titration will be used to evaluate the dose limiting (DLT) toxicity of each dose group, evaluate the safety and tolerance of Gentulizumab in the treatment of patients with progressive hematological malignancies, and determine the maximum tolerated dose (MTD) and phase II recommended dose (RP2D); At the same time, the pharmacokinetics (PK), pharmacodynamics (PD), immunogenicity, preliminary efficacy and biomarkers of gentulizumab will be evaluated to provide sufficient basis for new drug application (NDA) guidance and further clinical use.

DETAILED DESCRIPTION:
Gentulizumab, developed by GeneScience Pharmaceuticals Co., Ltd. has completed all non clinical related studies. The company applied for clinical trial in June 2020 (acceptance No.: CXSL2000164), and obtained the notice of approval of drug clinical trial (Notice No.: 2020LP00360) approved by National Medical Products Administration on September 3, 2020 to carry out clinical trial for hematological malignancies.

PD: Gentulizumab demonstrated the anticipated PD effects in corresponding tumor models in vitro and in vivo.

PK: The observed PK characteristics are consistent with other monoclonal antibodies.

Toxicology: In the toxicity test in cynomolgus monkeys after single-dosing and repeated dosing, reversible changes in erythroid indexes related to pharmacological action were observed. The MTD was 450 mg/kg and the NOAEL for repeat dosing was 300 mg/kg.

Safety Window: Based on results from the GLP-compliant 4-week repeat-dose toxicology study with 6-week recovery in cynomolgus monkeys (QW 5, i.v., 30, 100 or 300 mg/kg with a priming dose of 10 mg/kg), gentulizumab-related transient changes were noted in hematology, coagulation and clinical chemistry parameters and the NOAEL was determined to be 10+300 mg/kg. The human equivalent dose (HED) is 10+300 mg/kg converted based on body weight. The maximum recommended starting dose (MRSD) is considered to be 1.67+50 mg/kg (1/6 of HED of NOAEL) for advanced cancer treatment. The proposed human starting dose (0.1 mg/kg) provides a substantial safety margin, which is 16.7-500-fold lower than the MRSD and 100-3000-fold lower than the HED of NOAEL.

The trial is divided into 3 parts: priming dose exploration, therapeutic dose exploration and phase II recommended dose (RP2D) exploration.

The first part, priming dose exploration. In this part, 5 dose levels are planned. "3 + 3" dose escalation method combined with rapid titration will be adopted. Thirteen to Thirty subjects will be enrolled. The investigational drug is administered IV once a week and a dosing cycle is 4 weeks.

The study process of first three dose levels (0.03 mg/kg, 0.1 mg/kg, 0.3 mg/kg) of part one is shown below: screening period (4 weeks), observation period for dose limiting toxicity (4 weeks), continuous dosing period (once a week, until the discontinuation criteria are met), safety follow-up period after discontinuation (28 days after the last administration) and progression free survival follow-up period after discontinuation (once every 12 weeks until the survival follow-up endpoint). The study process of the last two dose levels (1 mg/kg, 3 mg/kg) is shown below: screening period (4 weeks), observation period for dose limiting toxicity (5 weeks including 1 week of single priming dose), continuous dosing period (once a week, until the discontinuation criteria are met), safety follow-up period after discontinuation (28 days after the last administration) and progression free survival follow-up period after discontinuation (once every 12 weeks until the survival follow-up endpoint).

Connection between part one and two.

Investigator and sponsor determine the optimal priming dose of part two together based on data from part one. The categories of data include:

1. The degree of abnormalities of the peripheral erythrocyte, white blood cell and platelet count.
2. Whether is there a compensatory increase in reticulocytes.
3. PD indicators (RO of red blood cells, white blood cells, platelets and tumor cells) If the conclusion of part one is "priming dose required", optimal priming dose will be determined and the dosing module of part two will be single optimal priming dose plus therapeutic dose escalation.

If the conclusion of part one is "priming dose not required", the dosing module of part two will be therapeutic dose escalation.

The second part, therapeutic dose exploration. The second part will be divided into 3 therapeutic dose levels (10 mg/kg, 30 mg/kg, 45 mg/kg). "3 + 3" dose escalation method will be adopted.

The number of subjects enrolled is 9-18. The investigational drug is administered IV once a week and a dosing cycle is 4 weeks.

The third part, exploration of RP2D As MTD is discovered during the second part, 6-10 subjects will be further enrolled at MTD level. More data of safety and tolerance will be acquired and used for the calculation of RP2D. The study process and administration method are the same as those in the second part.

Statistical analysis datasets Full analysis set (FAS): Based on the principle of intention-to-treat, all the subjects who are successfully enrolled and have at least one treatment record will be included in the full analysis set of this trial. The following situations may cause the enrolled subjects to be excluded from the FAS set: for example, they do not meet the primary inclusion criteria, they do not take the investigational drug once, they do not have any data after enrollment, etc. Demographic data, baseline data and efficacy indicator will be statistically analyzed based on FAS.

Safety analysis set (SS): include all the subjects who receive at least one treatment and have safety evaluation data after treatment. The safety population was primarily used for the analysis of safety data.

Pharmacokinetic data set (PKS): All subjects who were enrolled in the PKS and received at least one dose of the investigational drug and had PK evaluation data after administration constituted the PK analysis set of this study. In the PK analysis set, different PK parameters may include different numbers of subjects depending on the actual situation of trial completion.

ELIGIBILITY:
Inclusion Criteria:

1. The patient has the willingness to communicate with the Investigator, be able to understand and follow the trial requirements, volunteer to participate in the trial, understands and signs the written ICF, and is willing and able to comply with the visit schedule, administration plan, laboratory examination, and other clinical trial procedures.
2. Gender: Male or female.
3. Age ≥18
4. Life expectancy ≥ 3 months.
5. Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
6. Patients with relapsed/refractory AML or MDS for whom there exists no standard treatment options available.

   * AML diagnosed according to the 2016 WHO classification. Patients with acute promyelocytic leukemia (APL) are excluded. See Appendix 1.
   * For the patients MDS diagnosed according to the World Health Organization (WHO) classification system and evaluated as moderate-risk, high-risk, and very high-risk according to the Revised International Prognostic Scoring System (IPSS-R) for Myelodysplastic Syndrome.
7. The white blood cell (WBC) count in the patient's peripheral blood must be ≤ 20 × 109/L within 7 days of the first dose of the study drug. The patients with WBC count > 20 × 109/L may be treated with hydroxyurea (maximum dose 4 g/d) during the Screening period to achieve entry criteria. Hydroxyurea may be continued for the first 4 weeks of treatment (Cycle 1) to control blast counts at the discretion of the Investigator; hydroxyurea must be stopped after the first 4 weeks of treatment.
8. Hb levels must be above 5 g/dL on the day of the first dose of the study drug, and may be maintained by transfusion. Transfusion is permitted in the duration of trial.
9. Platelet count ≥ 10,000 cells/uL with no evidence of medically significant bleeding or medical predisposition to bleeding. Platelets may be maintained by transfusion at the discretion of the Investigator.
10. Adequate liver and kidney function as evidenced by meeting the following requirements:

    * Serum creatinine (Cr) ≤ 1.5 × the upper limit of normal (ULN) or creatinine clearance (CrCl) ≥ 60 mL/min (based on Cockcroft-Gault formula)
    * Aspartate aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN (≤ 5.0 times ULN for patients with liver metastasis/infiltration)
    * Serum total bilirubin (TBIL) ≤ 1.5 × ULN except for patients with Gilbert's syndrome, who are included if total bilirubin is < 3 × ULN or if direct bilirubin is < 1.5 × ULN.
11. Coagulation profile: prothrombin time (PT) ≤ 1.5 × ULN, international normalized ratio (INR) ≤ 1.5 × ULN or activated partial thromboplastin time (APTT) ≤ 1.5 × ULN.
12. Electrolytes and uric acid need to be stable and abnormalities correctable with medical intervention.
13. Patients must be willing to undergo bone marrow aspirates/biopsies per protocol specifications; these will be performed per protocol schedule to evaluate patient response to treatment.
14. Female patients with the possibility of pregnancy must consent to practice sexual abstinence or use of two highly effective forms of contraception, from the time of signing the ICF until at least 24 weeks after the end of dosing. Male patients with a partner of childbearing potential must consent to practice abstinence or use of two highly effective forms of contraception from the time of signing the ICF until at least 24 weeks after the end of dosing.

    * Note: Women who have undergone surgical sterilization (including hysterectomy, bilateral oophorectomy or total hysterectomy), or who are postmenopausal (defined as no menses for more than 12 consecutive months without medical interference) are considered to have no possibility of pregnancy.
15. Patients who have recovered from the toxic effects of the last treatment (CTCAE ≤ grade1, except for special circumstances such as alopecia, fatigue) before the first dosing, and whose corresponding AEs are judged by the Investigator as having no safety risks for treatment on the current study are eligible.

Exclusion Criteria:

1. Female patients who are pregnant or lactating or have a positive pregnancy test at baseline.
2. Patients with previous severe allergic reactions to the investigational drug or its components.
3. Patients who have received any of the following treatments:

   * Prior treatment with the CD47/SIRPα pathway as the therapeutic target.
   * Systemic antitumor therapy or any experimental therapy including within 7 days or 5 half-lives, whichever is longer, before the first dose. If a patient is receiving cytarabine, oral fluorouracils and endocrine therapy, the patient must be off the drug for at least 2 weeks or until the patient has recovered from toxic effects. If a patient is receiving nitrosourea, mitomycin or monoclonal antibody, the patient must be off the drug for at least 6 weeks or until the patient has recovered from toxic effects. If the elution time is insufficient due to schedule or PK characteristics, discussion with sponsor will be needed.
   * Expected to require treatment with other systemic anti-tumor therapies such as chemotherapy, immunotherapy, biotherapy or hormone therapy (except for palliative radiotherapy) during the study.
   * Prior vaccination with anti-tumor vaccines or live attenuated vaccines within 4 weeks before the first dosing.
   * Prior treatment with immunomodulatory drugs within 4 weeks before the first dose of study drug, except for topical, nasal and inhaled corticosteroids, or physiologic doses of systemic steroids (i.e., ≤ 10 mg/day prednisone or its equivalents).
4. Not Receiving any investigational drug within 4 weeks before the first administration, or participated in another clinical study at the same time except that the patient participated in an observational, non-intervention clinical study, or was in the follow-up period of an intervention clinical study.
5. No allogeneic transplantation within 6 months, no active graft-versus-host disease (GVHD), not receiving immunosuppressive treatment for GVHD within 4 weeks.
6. Symptomatic central nervous system metastases or primary leukemia including leptomeningeal disease or spinal cord compression. Patients with asymptomatic CNS disease who are radiologically and neurologically stable ≥ 4 weeks following CNS-directed therapy and are on a stable or decreasing dose of corticosteroids are eligible for study entry.
7. Patients with history of any active autoimmune disease, history of autoimmune disease, or disease or syndrome requiring treatment with systemic steroids or immunosuppressive medications (dermatological conditions that do not require systemic treatment or patients with resolved childhood asthma/allergies that do not require any intervention in adulthood; patients with a history of autoimmune-mediated hypothyroidism on a stable dose of thyroxine replacement therapy may be enrolled in the study).
8. History of immunodeficiency, including a positive HIV test, and other acquired, or congenital immunodeficiency disease.
9. History of ≥ Grade 3 thromboembolic event within the past 12 months, or current thrombolytic or anticoagulant therapy due to high risk of thrombus.
10. History of genetic or acquired causes of bleeding or anemia.
11. With cardiovascular diseases or manifestations including:

    * Congestive heart failure (NYHA class > 2).
    * History of unstable angina.
    * Myocardial infarction in the past 48 weeks.
    * Clinically significant malignant arrhythmia (excluding atrial fibrillation and paroxysmal supraventricular tachycardia unless hemodynamically significant).
    * Clinically significant QTcF prolongation (QTcF > 450 msec for males or QTcF > 470 msec for females).
    * Hypertension that cannot be well controlled (systolic blood pressure > 150 mmHg and diastolic blood pressure >80 mmHg), a history of hypertensive crisis, or a history of hypertensive encephalopathy.
12. Presence of active infection (fever that is felt to be caused by the tumor after work-up for infectious causes may be enrolled according to the judgment of the investigator).
13. Patients with active pulmonary tuberculosis infection confirmed by medical history or CT examination, or with a history of active pulmonary tuberculosis infection within 1 year before enrollment, or with a history of active pulmonary tuberculosis infection more than 1 year ago but without curative treatment.
14. Patients with active viral hepatitis B or C confirmed by serologic examinations, or defined as HBV-DNA > lower limit of detection or HCV-RNA > lower limit of detection when the conditions cannot be evaluated by serologic examinations (chronic hepatitis B or chronic hepatitis C can be treated with standardized antiviral therapy for stable disease).
15. Treponema pallidum antibody positive.
16. Major surgery or significant trauma within 4 weeks prior to the first dosing. Wound and injuries must be fully recovered.
17. Previous history of drug abuse, alcoholism, or drug addiction.
18. Concurrent malignancy within 2 years prior to entry other than adequately treated cervical carcinoma-in-situ, localized squamous cell cancer of the skin. The investigators expect both primary neoplasms could benefit from the study.
19. Patients with chronic obstructive pulmonary disease (COPD) or pulmonary fibrosis.
20. Any uncontrolled intercurrent illness or condition that in the judgment of the Investigator may endanger the patient.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2024-07-30 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
adverse events (AEs) | ICF signing to 90 days after last administration or initiation of new anti-tumor treatment
  Adverse events (AEs) refer to all adverse medical events occurred in subjects after the informed consent was signed, which may represent symptoms, signs, diseases, or laboratory examination abnormalities, but do not necessarily have a causal relationship with the investigational drug.
serious adverse events (SAEs) | ICF signing to 90 days after last administration or initiation of new anti-tumor treatment
  1. An SAE refers to any adverse medical event that meets any of the following criteria:
  2. Results in death
  3. Life-threatening: "Life-threatening" refers to an immediate risk of death for a severely ill patient and does not refer to the assumption that death may occur if it were to become severe in the future.
  4. Event resulting in hospitalization or prolongation of hospitalization.
  5. Event that results in significant or permanent disability/dysfunction. Disability refers to substantial disruption of a person's ability to perform normal activities of daily living.
  6. Results in a congenital anomaly or birth defect.
  7. Other important medical events: Events that may not immediately result in death, be life-threatening, or result in hospitalization/prolongation of hospitalization. However, based on medical judgment, these events may cause injuries to the subject or may require medical intervention to prevent any of the said circumstances from occurrence.

SECONDARY OUTCOMES:
The plasma drug peak concentration (Cmax) | First administration to 90 days after the last administration or initiation of new anti-tumor treatment
  Multiple dosing pharmacokinetic (PK) parameters
The area under the drug time curve (AUC) | First aAdministration to 90 days after the last administration or initiation of new anti-tumor treatment
  Multiple dosing pharmacokinetic (PK) parameters
Pharmacodynamic (PD) parameters | First administration to 90 days after the last administration or initiation of new anti-tumor treatment
  Receptor occupancy (RO) of gentulizumab of red blood cells, white blood cells, platelets and neoplastic cells in peripheral blood

OTHER OUTCOMES:
Anti-drug Antibody (ADA) and Neutralizing Antibody (NAb) | First administration to 28 days after the last administration or initiation of new anti-tumor treatment
Progression-free survival response) | From date that informed consent forms were signed until the date of disease progression
Duration of response response) | The duration from the first evaluation of the disease as complete response or partial response to the first evaluation as progressive disease or death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Junmin Li, Doctor, Principal Investigator — Ruijin Hospital
Locations (1):
- Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No